CLINICAL TRIAL: NCT06768216
Title: Effect of Indianized Version of Mediterranean Diet vs. Low Fat Diet on Hepatic Steatosis in Overweight Children and Adolescent With MASLD: A Randomized Control Trial
Brief Title: Effect of Indianized Version of Mediterranean Diet vs. Low Fat Diet on Hepatic Steatosis in Overweight Children and Adolescent With MASLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-MASDL-01
Record Dates: First submitted 2025-01-03; First posted 2025-01-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease
MeSH Terms: interventions — Diet, Fat-Restricted; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indianized version of Mediterranean Diet+Physical Activity (Active Comparator): Indo Mediterranean diet will have Carbohydrates 40-45%, fats 30-35% and proteins 15-20%. Mediterranean diet, it will be specified to use Mustard oil, use of specific fruits like orange, apple, mosambi (avoid high glycemic fruits), use more of green leafy vegetables, Use of multigrain atta (Home made- 10 kg of multigrain atta will have - 8 kg of wheat + 500g each of Ragi+Bajra+ Jowar + Chana dal flour). At least 45- 60 mins of exercise (peer group activity - cycling, football, brisk walking),
  Interventions: Other: Indianized version of Mediterranean Diet; Other: Physical Activity
- Low Fat Diet + Physical Activity (Experimental): Low fat diet will have 50-60% carbohydrate, 20-30% fat (with <10% saturated fat), and 20% protein. In the Low Fat Diet group, there will be only be restriction of total fat content to less than <30%. They can use whichever household oil, consume any fruit or vegetables, any atta and no restriction on diary or non-vegetarian diet.
  Interventions: Other: Low Fat Diet; Other: Physical Activity

INTERVENTIONS:
Other: Indianized version of Mediterranean Diet — Indo Mediterranean diet will have Carbohydrates 40-45%, fats 30-35% and proteins 15-20%. Mediterranean diet, it will be specified to use Mustard oil, use of specific fruits like orange, apple, mosambi (avoid high glycemic fruits), use more of green leafy vegetables, Use of multigrain atta (Home made- 10 kg of multigrain atta will have - 8 kg of wheat + 500g each of Ragi+Bajra+ Jowar + Chana dal flour).
  Arms: Indianized version of Mediterranean Diet+Physical Activity
Other: Low Fat Diet — Low fat diet will have 50-60% carbohydrate, 20-30% fat (with <10% saturated fat), and 20% protein. In the Low Fat Diet group, there will be only be restriction of total fat content to less than <30%. They can use whichever household oil, consume any fruit or vegetables, any atta and no restriction on diary or non-vegetarian diet. Along with this, both groups will be given a list of do's and dont's. In the list of Do's , it will be mentioned to Eat plenty of vegetables, Fruits, Nuts, Whole grains, Screen time of less <2 hrs /day (According to American academy of pediatrics) and Average hours of sleep in a day for age 8-18 = 8-9 hrs (According to American academy of sleep medicine). In the dont's list, it will be mentioned to avoid Sugar, Soda, Beverages, cold drinks, processed juices, processed food, junk foods, Maida, Ice cream, Creamy Desserts, Biscuit, chips and cake.
  Arms: Low Fat Diet + Physical Activity
Other: Physical Activity — At least 45- 60 mins of exercise (peer group activity - cycling, football, brisk walking),

SUMMARY:
NAFLD encompasses the entire spectrum of Fatty liver disease in individuals without significant alcohol consumption, ranging from fatty liver to steatohepatitis to cirrhosis. A high prevalence of NAFLD (62.5%) was observed in overweight/obese Indian adolescent (1). Lifestyle modification consisting of diet, exercise and weight loss has been advocated to treat patients with NAFLD (2). EASL guidelines recommends that the macronutrient in the diet should be adjusted according to the Mediterranean diet for weight loss (3). Mediterranean diet helps to decrease hepatic fat by decreasing lipogenesis, fibrogenesis, inflammation, oxidative stress and by increasing fatty acids beta oxidation (4). There are various studies showing benefits of using other diets such as Low Fat Diet, Low Carbdohydrate diet, Low Fructose Diet, et. Though there are numerous studies in adults comparing Mediterranean diet vs Low Fat diet, date regarding the same in children are lacking. The aim of this study will be to compare the Effect of Indianized version of Mediterranean diet vs. Low Fat Diet on Hepatic Steatosis in Overweight children and adolescent with MASLD.

DETAILED DESCRIPTION:
Aim: To Study the effect of Indianized version of Mediterranean diet versus Low Fat diet on Non-Invasive markers of hepatic steatosis in children and adolescent with MASLD.

Primary objective: To compare the proportions of patients achieving normal CAP values (<236db/m) after 180 days of IMD versus LFD in children and adolescent with MASLD.

Secondary objectives:

* To compare the changes in CAP values after 180 days of IMD versus LFD in children and adolescent with MASLD.
* To compare the grades of Fatty liver on Ultrasonography after 180 days between the two study groups.
* To compare the changes in CAP value in PNPLA3 mutant children.
* To study the change in Adiponectin, Cytokines(TNF alpha, IL 6, IL-1β, and IL-17) after 180 days between the two study groups.
* To compare the changes in following parameters in both study groups: Weight, BMI, HOMA IR and Lipid profile.
* To compare the adherence to IMD, with the help of Modified KIDMED score.
* Study design: Prospective, Randomized, Single center Open label study.
* Children and adolescent aged 8 to 18 years with CAP > 236dB/m will be enrolled in the study. Consent for dietary intervention will be taken. Baseline parameters analysed includes:

  * Anthropometry :

    - Weight, Height, BMI, Waist circumference
  * Imaging:

    - Ultrasonography abdomen, Fibroscan (LSM, CAP values)
  * Biochemical parameters:

    - ALT, AST, Lipid profile, HOMA IR
  * Adiponectin & Cytokines: TNF alpha, IL6, IL-1β, and IL-17
  * Liver Biopsy when indicated: ALT>80, LSM>8.6.
* Intervention:

Both the groups will have be given a handmade individualised (according to weight) specific diet to follow. Indo-Mediterranean diet will be given to one group and other group will have Calorie restricted diet. Indo Mediterranean diet will have Carbohydrates 40-45%, fats 30-35% and proteins 15-20%. Low fat diet will have 50-60% carbohydrate, 20-30% fat (with <10% saturated fat), and 20% protein. Calories will be calculated according to the age specified RDA from ICMR guidelines. In Indo-Mediterranean diet, it will be specified to use Mustard oil, use of specific fruits like orange, apple, mosambi (avoid high glycemic fruits), use more of green leafy vegetables, Use of multigrain atta (Home made- 10 kg of multigrain atta will have - 8 kg of wheat + 500g each of Ragi+Bajra+ Jowar + Chana dal flour). They will be advised to eat Dairy products in moderation and if non vegetarian diet (Fish, chicken, only twice a week). Dry fruits (Walnuts) and herbs (cinnamon, garlic, basil, and pepper) will be an important part of the diet. In the Low Fat Diet group, there will be only be restriction of total fat content to less than <30%. They can use whichever household oil, consume any fruit or vegetables, any atta and no restriction on diary or non-vegetarian diet. Along with this, both groups will be given a list of do's and dont's. In the list of Do's , it will be mentioned to Eat plenty of vegetables, Fruits, Nuts, Whole grains, at least 45- 60 mins of exercise (peer group activity - cycling, football, brisk walking), Screen time of less <2 hrs /day (According to American academy of pediatrics) and Average hours of sleep in a day for age 8-18 = 8-9 hrs (According to American academy of sleep medicine). In the dont's list, it will be mentioned to avoid Sugar, Soda, Beverages, cold drinks, processed juices, processed food, junk foods, Maida, Ice cream, Creamy Desserts, Biscuit, chips and cake.

• Monitoring and assessment: All Parameters will be re-assessed at 180 days (except liver biopsy). Both groups will be explained to maintain a food diary mentioning cheat days (Food other than the diet given), screen time (<2hrs/day), Exercise (45-60 mins/day, parameters will be checked by pedometer app) and average hours of sleep (8-9hrs/day). Food diary will be checked once in two weeks on phone calls or virtual OPD. Once weekly phone calls (30 mins) will be checked to see the adherence and to motivate the child. They will be required to follow up in OPD once in a month. Adherence to Indo Mediterranean diet will be assessed by Modified KIDMED score.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 8-18 years
2. BMI > 85th centile
3. CAP > 236

Exclusion Criteria:

- Other Liver diseases such as Viral hepatitis (Hep B and C), Autoimmune hepatitis, Wilson disease.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the proportions of patients achieving normal CAP values (<236db/m) after 180 days of IMD versus LFD in children and adolescent with MASLD. | 180 days

SECONDARY OUTCOMES:
To compare the changes in CAP values after 180 days of IMD versus LFD in children and adolescent with MASLD. | 180 days
To compare the grades of Fatty liver on Ultrasonography after 180 days between the two study groups. | 180 days
To compare the changes in CAP value in PNPLA3 mutant children. | 180 days
To study the change in Adiponectin, Cytokines(TNF alpha, IL 6, IL-1β, and IL-17) after 180 days between the two study groups. | 180 days
To compare the changes in following parameters in both study groups: Weight. | 180 days
To compare the changes in following parameters in both study groups: BMI. | 180 days
To compare the changes in following parameters in both study groups: HOMA IR . | 180 days
To compare the changes in following parameters in both study groups: Lipid profile. | 180 days
To compare the adherence to IMD, with the help of Modified KIDMED score. | 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided